CLINICAL TRIAL: NCT06886438
Title: Comparison of Regenerative Endodontic Procedures Using Periapical Bleeding Induction, L-PRF, and I-PRF in Mature Teeth With Periapical Lesions: A Randomized Controlled Clinical Trial
Brief Title: Periapical Bleeding Versus PRF Techniques in Regenerative Endodontic Therapy: A Randomized Controlled Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Saglik Bilimleri Universitesi (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HKORUCU1; 2023/056 (Other Grant/Funding Number: Scientific Research Projects Coordination Unit of Health Sciences University)
Record Dates: First submitted 2025-02-13; First posted 2025-03-20 (Actual); Last update posted 2025-03-20 (Actual); Status verified 2025-01

CONDITIONS: Necrotic Pulp; Regenerative Endodontic Procedures; Mature Teeth; Apical Periodontitis; PRF; Discoloration of Teeth
MeSH Terms: conditions — Dental Pulp Necrosis; Periapical Periodontitis; Tooth Discoloration

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- AP (Experimental): Necrotic pulped, mature teeth with apical periodontitis.
  Interventions: Procedure: RVS; Procedure: L-PRF; Procedure: i-PRF

INTERVENTIONS:
Procedure: RVS — Revascularization
Procedure: L-PRF — Regenerative endodontic procedure with L-PRF application
Procedure: i-PRF — Regenerative endodontic procedure with i-PRF application

SUMMARY:
This study investigates a biological approach that allows infected and necrotic teeth to heal themselves instead of being treated with traditional root canal therapy. Traditional root canal treatment involves cleaning the infected tissue inside the tooth and sealing it with a filling material, whereas regenerative endodontic treatment is a novel approach that enables the tooth to repair itself. This treatment method involves inducing bleeding in the root area or applying special blood derivatives (PRF types) to accumulate healing-supporting cells and growth factors. The aim of the study is to compare the effects of different biological treatment methods on the healing process, postoperative pain, and tooth discoloration. The results may help develop more effective and aesthetically successful treatment options in the future.

DETAILED DESCRIPTION:
This study investigates the effectiveness of regenerative endodontic procedures in the treatment of necrotic and infected teeth. Traditional root canal treatment involves the complete removal of infected tissue from inside the tooth and sealing the root canal with a biocompatible filling material. However, this method does not restore the tooth's natural vitality or protective mechanisms. Additionally, it may increase tooth fragility and lead to discoloration over time.

Regenerative endodontic treatment is a biological approach that promotes the self-healing of the tooth. This method applies tissue engineering principles to stimulate the formation of new tissue within the root canal. During the treatment process, either bleeding is induced at the root tip or special platelet-rich fibrin (PRF) derivatives are applied to facilitate the accumulation of stem cells, growth factors, and immune-boosting components that support healing.

This study compares the effects of different regenerative treatment methods (bleeding induction, L-PRF, and I-PRF applications) on lesion healing, postoperative pain, and tooth discoloration. By determining the most effective method for teeth with completed root development and apical lesions, the study aims to establish an optimal treatment protocol for clinical practice. The findings will contribute to the development of treatment options that preserve the natural structure of the tooth, enhance aesthetics, and improve patient comfort and long-term treatment success.

ELIGIBILITY:
Inclusion Criteria:

* Single-rooted teeth with mature teeth with necrotic pulp requiring endodontic treatment, and a periapical lesion (Periapical Index Score (PAI) ≥3).
* Individuals without systemic diseases, not using antibiotics, corticosteroids, antidiabetic, or antihypertensive medications, and not pregnant.
* Patients without acute pain.
* Patients without extraoral swelling, sinus tract, or acute apical abscess.
* Individuals willing to participate and able to attend follow-up sessions regularly.

Exclusion Criteria:

* Teeth with internal or external root resorption or vertical root fractures.
* Immature teeth.
* Individuals outside the age range of 14-65 years.
* Patients with complicated systemic diseases or those using antibiotics, corticosteroids, antidiabetic, or antihypertensive medications.
* Patients with acute pain, those who have taken analgesic medication in the last 24 hours, or those who have used antibiotics within two weeks before treatment.
* Patients who are unlikely to attend follow-up sessions.

Ages: 14 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2024-02-03 (Actual); Primary Completion 2024-03-10 (Actual); Study Completion 2025-01-24 (Actual)

PRIMARY OUTCOMES:
Radiographic Assessment of Lesion Healing at 6 Months | Baseline and 6 months
  Lesion healing will be evaluated using periapical radiographs with the parallel technique, and the Periapical Index (PAI) will be used for the assessment of lesion healing.
Change in Pain Level at 24 Hours, 72 Hours, and 1 Week Post-Treatment | Post-Treatment at 24 Hours, 72 Hours, and 1 Week
  Pain levels will be assessed using the Numerical Rating Scale (NRS), ranging from 0 (no pain) to 100 (worst pain), measured at 24 hours, 72 hours, and 1 week post-procedure.
Assessment of Tooth Discoloration at 6 Months | Baseline and 6 months
  Tooth discoloration will be evaluated using a spectrophotometer based on the CIELab system, and teeth with a ΔE value greater than 3 will be considered discolored.

CONTACTS AND LOCATIONS:
Locations (1):
- Gulhane Faculty of Dentistry, University of Health Sciences, Ankara, Etlik, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
The impact of gender differences on pain assessment in the study was also evaluated. Additionally, the effect of age on lesion healing was analyzed. Since the study examines the effects of demographic data on lesion healing and post-treatment pain, demographic data will be shared.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code